CLINICAL TRIAL: NCT05467917
Title: ARMOR-Household: Characterizing Transmission of COVID-19 in Households of Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) Index Cases
Brief Title: ARMOR-Household: Characterizing Transmission of COVID-19 in Households of SARS-CoV-2 Index Cases
Status: Active, not recruiting | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: AAAS9688
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: COVID-19; Households; SARS CoV 2 Infection
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional genetic testing will be performed on saliva and cells collected from the participant's and household's swab, saliva, and blood.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Index Case: a) minor testing positive for SARS-CoV-2; b) symptomatic health workers or any individual with a history of exposure to SARS-CoV-2 confirmed positive patients; c) health workers or any individual who tests positive regardless of symptoms. Index case must be living in a multi-person household that includes at least one child with a history of exposure to SARS-CoV-2 positive patients
- Household Contact: Anyone residing in the house for at least 24 hours at the time of the index case diagnosis or study enrollment.

SUMMARY:
The goal of this project is to understand the household level transmission dynamics and factors that predict transmission of SARS-COV-2 between pediatric and adults in the household.

The novel coronavirus SARS-CoV-2 has spread all around the world and testing has posed a challenge globally. Not much is known about who does and does not acquire SARS-CoV2. It is also unknown who will show symptoms or progress severe disease or death from COVID-19. Children tend to have milder symptoms or none at all. Therefore, few children have ever been tested, so it is unknown if they get the infection as much as anyone else. Health care providers are highly exposed, and they do not get tested unless they show severe symptoms. If groups like children and health workers are infected, they can unknowingly spread SARS-CoV-2, unless they practice behaviors like self-isolation very strictly. The investigators aim to measure the prevalence of SARS-CoV-2 in children and health care workers at a large urban health center. The investigators will also measure how many people in the household of the positive children and health care workers also get SARS-CoV-2 infection. Lastly, the investigators will see what other risk factors affect who acquires SARSCoV-2 from inside or outside of the household clusters.

DETAILED DESCRIPTION:
The rapid spread of the novel coronavirus SARS-CoV-2 has resulted in pandemic levels and a global challenge in diagnosing infection. Little is known about transmission and disease presentation of COVID-19. Children tend to present with mild or no symptoms, and only a minority seem to progress to severe disease. Therefore, fewer have been tested. Health care providers who are highly exposed are under tested for their level of exposure. Under diagnoses in these groups can result in onward transmission of SARS-CoV-2 if non-pharmaceutical interventions like self-isolation are not strictly practiced. The investigators aim to assess the prevalence of SARS-CoV-2 in a pediatric, health care worker and other individuals sample in a large urban health center; Estimate the household secondary attack rate of SARS-COV-2 from the pediatric and adult index case SARS-COV-2 identified through the prevalence survey; and identify risk factors that affect transmission from within and outside of the household clusters.

This is an observational prospective cohort study of pediatric patients, New York Presbyterian (and affiliates) health workers, and any individuals who have been exposed to SARS-CoV-2 cases and their household contacts residing in New York City. Child index and their household members who consent to participate will be enrolled and tested for SARS-CoV-2. Households will be followed prospectively for a minimum of 15 days from the date the last household member testing positive. Daily clinical symptom reporting, social distancing behaviors within and outside of the household, emotional and mental health factors such anxiety, stigma and disclosure (among SARS-CoV-2 diagnosed) will be reported by adult household members and minors over the age of 7. Adults will report signs and symptoms for minors under the age of 7. SARS-CoV-2 negative household members will be re-tested around the day of onset of symptoms and baseline negative household members will be tested at the end of the observation period. A proportion of SARS-CoV-2 positive household members will be sampled serially for viral shedding and would be sampled on the day of onset of exposure. Households where all members are positive at baseline visit will be excluded from participation.

ELIGIBILITY:
Inclusion Criteria:

* Index is a positive child AND at least one household member is negative

OR

* Index is a positive symptomatic / asymptomatic New York Presbyterian Hospital (NYP) and affiliates worker or any individual AND at least one household member is negative

OR

* Either Index case is negative, exposed to a confirmed positive SARS-CoV-2 case, AND at least one household members is negative

Exclusion Criteria:

* Index case is positive and all household members are positive

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pediatric patients, New York Presbyterian health workers, and any individual who has been exposed to SARS-CoV-2 cases and their household contacts residing in New York City.
Sampling Method: Non-Probability Sample
Enrollment: 374 (Estimated)
Dates: Start 2021-08-01 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Period prevalence of SARS-CoV-2 Infection | Up to 28 days
  Period prevalence of SARS-CoV-2 infection as detected by use of home nasal swab and blood samples. At home nasal swab every 48-72 hours for about 15 days, with another potential collection on day 21 and day 28 of the study. Blood sample collected at enrollment and at day 28.
Household secondary attack rate of SARS-COV-2 | Up to 28 Days
  Household secondary attack rate of SARS-COV-2 from the pediatric and adult index case SARS-COV-2 identified through the prevalence survey in outcome 1. SARS-CoV-2 negative household members will be re-tested around the day of onset of symptoms and baseline negative household members will be tested at the end of the observation period. A proportion of SARS-CoV-2 positive household members will be sampled serially for viral shedding and would be sampled on the day of onset of exposure.
Identify risk factors associated within and extra-household transmission of SARS-CoV-2 | Up to 28 Days
  Identify sociodemographic, behavioral (e.g., social distancing behaviors within and outside of the household), clinical, and viral risk factors associated within and extra-household transmission of SARS-CoV-2 overall and by type of index cases. Daily clinical symptom reporting, social distancing behaviors within and outside of the household, emotional and mental health factors such anxiety, stigma and disclosure (among SARS-CoV-2 diagnosed) will be reported by adult household members and minors over the age of 7.

CONTACTS AND LOCATIONS:
Overall Officials: Delivette Castor, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Irving Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No